CLINICAL TRIAL: NCT02372461
Title: A Double Blind Community-based Randomized Trial of Amoxicillin Versus Placebo for Fast Breathing Pneumonia in Children Aged 2-59 Months in Karachi, Pakistan
Brief Title: Randomized Trial of Amoxicillin Versus Placebo for (Fast Breathing) Pneumonia
Acronym: RETAPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dr Fyezah Jehan, Associate Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MR/L004283/1; OPP1158281 (Other Grant/Funding Number: Bill & Melinda Gates Foundation)
Record Dates: First submitted 2014-11-04; First posted 2015-02-26 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Pneumonia; Tachypnea
Keywords: Amoxicillin; Placebo
MeSH Terms: conditions — Pneumonia; Tachypnea | interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Control (Active Comparator): Amoxicillin Liquid
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Placebo — This is an non inferiority trial, the intervention is a placebo
  Arms: Experimental
Drug: Amoxicillin — Amoxicillin Liquid
  Arms: Control

SUMMARY:
The relative benefits and risks of antibiotic therapy in WHO defined fast breathing pneumonia in pre-school children in resource limited settings are controversial both at an individual and public health level. Most infections are viral or self-limiting and non-selective drug treatment has contributed to the global epidemic of antibiotic resistance. There is no high quality trial evidence in managing children with fast breathing in community settings and the WHO itself has called for evidence on which to update guidance. The investigators proposed non inferiority trial comparing standard antibiotic treatment with placebo in poor urban slum settings in South Asia to address this deficit.

DETAILED DESCRIPTION:
Pneumonia is a major cause of illness and death in children in low-income countries. With a view to decreasing death from pneumonia, the World Health Organization and UNICEF developed the Integrated Management of Childhood Illness (IMCI) algorithm which simplifies management of common childhood illnesses such as pneumonia and diarrhea into different levels of severity for determining the most appropriate case management by primary healthcare providers. Many pneumonia cases are categorized as non-severe pneumonia (defined as fast breathing above the specified age cut-off for respiratory rates). As there is incomplete information regarding the cause of this type of "pneumonia" from primary care settings, treatment guidelines by WHO are dictated by culture information from hospital pneumonia cases which are different in severity and cause. Current WHO guidelines advocate the use of oral antibiotics for fast breathing pneumonia. However, it is postulated that most fast breathing pneumonia not requiring hospitalization is of viral etiology, thus does not require antibiotic treatment. The cost of antibiotic treatment for all children with pneumonia is high; an estimated US$ 200 million in South Asia & sub Saharan Africa alone. Since more than 60% of pneumonia is classified as non-severe (fast breathing), this puts a strain on already under-sourced programmes in low-income countries. Giving antibiotics where they confer no benefit also puts the child at risk of side effects and increases the risk of antimicrobial resistance in the community. This uncertainty forms the basis of the proposed study. Investigators propose to show in a clinical trial that the outcome of children diagnosed with WHO defined fast breathing pneumonia is similar regardless of whether they receive antibiotics or not. This study will be conducted in five primary health care centers located in low income communities of Karachi, Pakistan, with extensive trial experience. Children identified to have fast breathing without any danger signs will be randomized to receive either three days of the WHO recommended oral antibiotic (amoxicillin 250mg/5ml using WHO weight bands) or matching placebo (a drug that will taste and look like the amoxicillin but will not have an active ingredient) by a study physician working at the primary health center. The assignment of the antibiotic amoxicillin or placebo to a child will be done using a computer generated randomization list in a manner that at the end of the trial, there are equal numbers of children in both arms of the trial. Based on the statistical calculations for sample size, investigators need to assign 1214 children to receive amoxicillin and the same number of children to receive placebo. All children will receive the antibiotic or placebo under supervision of the primary health care physician in the morning. Evening doses will be delivered by locally hired Community Health Workers (CHWs) visiting the children at their home. All children will be assessed again on day 3 by a study physician to see if the child's presenting sign of high respiratory rate has resolved or not. All children with persistently high respiratory rate and/or development of a new clinical sign indicating illness progression will be labeled a treatment failure. There will invariably be some children with treatment failure in both the treatment arms; investigators hypothesize that there will be equal number of treatment failures in both the groups i.e. around 5%.

ELIGIBILITY:
Inclusion Criteria:

* History of cough or difficult breathing < 14 days (observed or reported) AND
* Respiratory rate ≥ 50 breaths per minute in children 2 to <12 months (on two consecutive readings by independent physicians) OR respiratory rate ≥ 40 breaths per minute in children12- 59 months (on two consecutive readings by independent physicians) AND
* Written informed consent by a legal guardian

Exclusion Criteria:

* Previously enrolled in study
* Pedal edema
* History of hospitalization in last two weeks
* With severe lower chest wall in-drawing
* Known asthmatics,TB or other severe illness
* Antibiotics taken in last 48 hours
* Bulging fontanel
* Congenital heart disease
* Any surgical condition requiring hospitalization
* Out of catchment area
* Any general danger sign as defined by WHO: Stridor when calm; hypoxia (SaO2 < 90% in air) ; inability to feed; persistent vomiting (after three attempts to feed the baby within ½ hour); convulsions; reduced conscious level

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4000 (Actual)
Dates: Start 2014-11-09 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Cumulative Treatment failure | Day 0-3
  Primary outcome will be cumulative treatment failure at or before 3 days. The following definitions will be used: either death, any danger sign, onset of chest in drawing as defined by WHO, hospitalization due to any reason, change in antibiotic regimen by study physician for new-onset infectious co-morbidity or change in antibiotic regimen by study physician for serious non-fatal antibiotic-associated adverse event on or before day 3.

SECONDARY OUTCOMES:
Relapse | Day 4-14
  Same definition as treatment failure but during Day 4-14

CONTACTS AND LOCATIONS:
Overall Officials: Fyezah Jehan, Msc, Principal Investigator — Aga Khan Univeristy
Locations (1):
- PHC at Ibrahim Haidry Goth, Ali Akber Shah Colony, Rerhi Goth, Bhains Colony, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jehan F, Nisar I, Kerai S, Balouch B, Brown N, Rahman N, Rizvi A, Shafiq Y, Zaidi AKM. Randomized Trial of Amoxicillin for Pneumonia in Pakistan. N Engl J Med. 2020 Jul 2;383(1):24-34. doi: 10.1056/NEJMoa1911998. PMID 32609980
- [Derived] Brown N, Rizvi A, Kerai S, Nisar MI, Rahman N, Baloch B, Jehan F. Recurrence of WHO-defined fast breathing pneumonia among infants, its occurrence and predictors in Pakistan: a nested case-control analysis. BMJ Open. 2020 Jan 7;10(1):e035277. doi: 10.1136/bmjopen-2019-035277. PMID 31915178
- [Derived] Jehan F, Nisar MI, Kerai S, Brown N, Balouch B, Hyder Z, Ambler G, Ginsburg AS, Zaidi AK. A double blind community-based randomized trial of amoxicillin versus placebo for fast breathing pneumonia in children aged 2-59 months in Karachi, Pakistan (RETAPP). BMC Infect Dis. 2016 Jan 13;16:13. doi: 10.1186/s12879-015-1334-9. PMID 26758747